CLINICAL TRIAL: NCT05898724
Title: Assessment of the Rate of Oseointegration Surrounding Nano-coated Orthodontic Titanium Miniscrew
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud M. Fathy Aboelmahasen, Lecture of orthodontics - Faculty of dental medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 915/307
Record Dates: First submitted 2023-05-09; First posted 2023-06-12 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Health Care Utilization; Diet, Healthy; Frey Syndrome
MeSH Terms: conditions — Patient Acceptance of Health Care; Sweating, Gustatory | interventions — Zinc Oxide

STUDY DESIGN:
Intervention Model Description: The present study will include 18 Egyptian males orthodontic patients divided into three groups; blank group, silver hydroxyapatite group, zinc oxide group. Each group will include six patients that will have a surgical procedure to install two orthodontic miniscrews (blank or nano-coated) (1.6 mm diameter and 6 mm length).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Blank group (Experimental): Blank group: include six orthodontic patients, which have a surgical procedure to install two orthodontic titanium miniscrews in the two lateral parts of the maxilla of each patient, so this group will include 12 installed orthodontic titanium miniscrews.
  Interventions: Procedure: Blank group
- Silver hydroxyapatite group: (Experimental): Silver hydroxyapatite group: include six orthodontic patients, which have a surgical procedure to install two silver hydroxyapatite nano-coated orthodontic titanium miniscrews in the two lateral parts of the maxilla of each patient, so this group will include 12 installed silver hydroxyapatite nano-coated orthodontic titanium miniscrews.
  Interventions: Procedure: Silver hydroxyapatite
- Zinc oxide group (Experimental): Zinc oxide group: include six orthodontic patients, which have a surgical procedure to install two zinc oxide nano-coated orthodontic titanium miniscrews in the two lateral parts of the maxilla of each patient, so this group will include 12 installed zinc oxide nano-coated orthodontic titanium miniscrews.
  Interventions: Procedure: Zinc oxide

INTERVENTIONS:
Procedure: Blank group — include six orthodontic patients, which have a surgical procedure to install two orthodontic titanium miniscrews in the two lateral parts of the maxilla of each patient, so this group will include 12 installed orthodontic titanium miniscrews.
  Arms: Blank group
Procedure: Silver hydroxyapatite — include six orthodontic patients, which have a surgical procedure to install two silver hydroxyapatite nano-coated orthodontic titanium miniscrews in the two lateral parts of the maxilla of each patient, so this group will include 12 installed silver hydroxyapatite nano-coated orthodontic titanium miniscrews.
  Arms: Silver hydroxyapatite group:
Procedure: Zinc oxide — include six orthodontic patients, which have a surgical procedure to install two zinc oxide nano-coated orthodontic titanium miniscrews in the two lateral parts of the maxilla of each patient, so this group will include 12 installed zinc oxide nano-coated orthodontic titanium miniscrews.
  Arms: Zinc oxide group

SUMMARY:
The current study was directed to evaluate rate of oseointegration surrounding nano-coated orthodontic titanium miniscrew.The current study will conduct on eighteen Egyptian males orthodontic patients for three months.

Study Groups:

A- Blank group: include six orthodontic patients, which have a surgical procedure to install two orthodontic titanium miniscrews in the two lateral parts of the maxilla , so this group will include 12 installed orthodontic titanium miniscrews.

B- Silver hydroxyapatite group: include six orthodontic patients, which have a surgical procedure to install two silver hydroxyapatite nano-coated orthodontic titanium miniscrews in the two lateral parts of the maxilla, so this group will include 12 installed silver hydroxyapatite nano-coated orthodontic titanium miniscrews.

C- Zinc oxide group: include six orthodontic patients, which have a surgical procedure to install two zinc oxide nano-coated orthodontic titanium miniscrews in the two lateral parts of the maxilla, so this group will include 12 installed zinc oxide nano-coated orthodontic titanium miniscrews.

DETAILED DESCRIPTION:
The present study will include 18 Egyptian males orthodontic patients divided into three groups; blank group, silver hydroxyapatite group, zinc oxide group. Each group will include six orthodontic patients that will have a surgical procedure to install two orthodontic miniscrews (blank or nano-coated) (1.6 mm diameter and 6 mm length). The Surgical procedure in all groups will performed by the same operator.

Before installation of the orthodontic miniscrews, each participant should have local anesthesia . The two orthodontic miniscrews will install in the two lateral parts of anterior maxilla; one in the right side and another in the left side. The orthodontic miniscrews (The Tomas® orthodontic mini-screws will purchase from Dentaurum Company (Germany) and will be placed by specific driver perpendicular on the installed surface (90 degree).

The head of the orthodontic miniscrews that will use in the current study (blank or nano-coated) will be coated by 3 mm dental composite resin (Z fill, 3M ESPE, St. Paul, MN, USA) to prevent transferring of any heat to the tissues that surround the orthodontic miniscrew and so this may affect the partial oseointegration and stability of the orthodontic miniscrews.

Assessment of quality and quantity of oseointegration.

For assessment of quality and quantity of oseointegration, each orthodontic patient have a CBCT (Cone beam computed tomography) that will take by using Planmeca Romexis MD 3D Extraoral Imaging System. CBCT datasets were acquired by software with reconstruction slice thickness of 0.2 mm and 728 X 728 matrix. The CBCT was made by high resolution scan that was made with isotropic voxel size set at 200mm and 10 X 15 cm field of view. The raw images were exported into Digital Imaging and Communications in Medicine (DICOM). All landmark identifications and measurements were made using Planmeca Romexis Viewer 4.4.2.R 3D Imaging Software. The CBCT will be taken just after installation of the orthodontic miniscrews and after three months of installation.

ELIGIBILITY:
Inclusion Criteria:

1. Health Care Utilization.
2. Daily high calcium meals.
3. free from any systemic diseases.
4. Oral cavity is free from any injury or ulcers

Exclusion Criteria:

1. systemic diseases.
2. fracture of the jaw.
3. injuries or ulcers within the oral cavity

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The current study will conduct on eighteen Egyptian males.
Enrollment: 18 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
assessment of quality of oseointegration | three months
  each patient have a CBCT (Cone beam computed tomography) that will take by using Planmeca Romexis MD 3D Extraoral Imaging System. CBCT datasets were acquired by software with reconstruction slice thickness of 0.2 mm and 728 X 728 matrix. The CBCT was made by high resolution scan that was made with isotropic voxel size set at 200mm and 10 X 15 cm field of view. The raw images were exported into Digital Imaging and Communications in Medicine (DICOM). All landmark identifications and measurements were made using Planmeca Romexis Viewer 4.4.2.R 3D Imaging Software. The CBCT will be taken just after installation of the orthodontic miniscrews and after three months of installation.

SECONDARY OUTCOMES:
Microbial interaction | three months
  by taking 18 swabs from oral cavity surround each orthodontic mini-screw (blank, silver hydroxyapatite, zinc oxide), after that the swab is analysed to assess the microbial action against normal flora of the oral cavity of the the orthodontic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud MF Abo - Elmahasen, PHD, Principal Investigator — Lecturer of orthodontics - Faculty of dental medicine - Al-Azhar university
Locations (1):
- Nasr city, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No